CLINICAL TRIAL: NCT01808261
Title: Study MAG104615, a Proof of Concept Study for GSK249320 Versus Placebo in Stroke Patients
Brief Title: Proof of Concept (POC) in Patients With Ischaemic Stroke
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated for futility.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 104615
Record Dates: First submitted 2013-02-14; First posted 2013-03-11 (Estimated); Results first posted 2017-10-03 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-09

CONDITIONS: Cerebrovascular Accident
Keywords: Ischemic Stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo is a clear, colorless solution (50mM acetate buffer, pH 5.5 containing 0.02% (w/v) polysorbate-80 and made isotonic with 111.2 mM sodium chloride). Placebo is for intravenous (IV) use only.
  Interventions: Drug: Placebo
- GSK249320 100/mg (Active Comparator): Clear to opalescent, colorless to pale yellow or pale brown, and is supplied as a sterile, concentrated solution (1000mg/vial). GSK249320 is for IV use only.
  Interventions: Drug: GSK249320 100/mg

INTERVENTIONS:
Drug: GSK249320 100/mg — Clear to opalescent, colorless to pale yellow or pale brown, and is supplied as a sterile, concentrated solution (1000mg/vial). GSK249320 is for IV use only.
  Arms: GSK249320 100/mg
Drug: Placebo — Placebo is a clear, colorless solution (50mM acetate buffer, pH 5.5 containing 0.02% (w/v) polysorbate-80 and made isotonic with 111.2 mM sodium chloride). Placebo is for intravenous (IV) use only.
  Arms: Placebo

SUMMARY:
Study MAG104615, a Proof of Concept Study for GSK249320 versus placebo in Stroke Patients.

DETAILED DESCRIPTION:
Myelin-associated glycoprotein (MAG) is one of the key proteins known to inhibit neuronal regeneration when released from oligodendrocytes in conditions of neuronal injury, such as stroke. GSK249320 is a humanised monoclonal antibody (mAb) that binds with high specificity to MAG and antagonises or neutralises MAG-mediated inhibition and has been shown to improve functional recovery after stroke in pre-clinical models, possibly by promoting neuroregeneration and plasticity. The present study (MAG104615) is designed to establish Proof of Concept (PoC) for GSK249320 in ischemic stroke patients. MAG104615 will be a placebo-controlled, double-blind, multicenter, randomized, repeat dose, Bayesian design study. PoC will be achieved by demonstrating a clinically meaningful improvement in lower limb motor recovery, specifically by evaluating changes in gait velocity from baseline to Day 90/Month 3. Subjects will also be followed out to Day 180/Month 6 to further evaluate longer term motor recovery and safety. Additional secondary efficacy measures of motor recovery will be evaluated to further demonstrate and characterize the extent and duration of overall motor recovery after treatment with GSK249320. Changes in disability and neurological impairment will be characterized after treatment with GSK249320 and explored for how they relate to motor recovery. This PoC study will also further characterize the safety, PK, and immunogenicity of GSK249320 will explore pharmacodynamic (PD) markers, and will explore use of actigraphy to measure motor recovery. Subjects will be stratified by gait velocity at baseline for randomization (1:1 allocation) into one of two treatment groups: 15mg/kg GSK249320, or placebo. Each subject will receive 2 repeat IV doses of GSK249320 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed diagnosis of stroke according to the World Health Organization definition which is, 'a rapid onset event of vascular origin reflecting a focal disturbance of cerebral function, excluding isolated impairments of higher function, and persisting longer than 24 hours [World Health Organization, 1989].
* Stroke onset must be within the last 24-72 hours of the first infusion of Investigational Product. Time of stroke onset is defined at the time at which the patient/relative is first aware of the stroke deficit. For patients who awake with deficits, or who are found unconscious, the time of onset is defined as the time at which they were last known to be symptom free.
* Have a stroke that is radiologically confirmed to be ischemic and supratentorial. The diameter of the ischemic lesion is >15mm in any single direction or the volume is >4cc. See the Study Procedures Manual (SPM) for guidance on how to calculate the lesion size.
* Have a total NIHSS score of 3-21.
* Have a lower limb deficit from the incident stroke which is defined as a score of 1-4 on the NIHSS Motor Leg question (question #6).
* Aged 18-90, inclusive.
* Expectation the subject will receive standard physical, occupational and speech rehabilitation therapy as indicated for the post stroke deficits.
* Male subjects and female subjects of non-child-bearing and child-bearing potential are allowed to participate in this study. See Section 11, Appendix 1 for definitions. Females of child-bearing potential must have a negative pregnancy test prior to enrollment and must agree to use one of the contraceptive methods specified in Section 11, Appendix 1.

Exclusion Criteria:

* Ability to walk >0.8m/s as measured by the Gait Velocity assessment.
* History of a previous symptomatic stroke within 3 months prior to study entry.
* Presence of significant disability prior to the current stroke. Significant disability is defined as having a pre-stroke Rankin score of >2.
* Subjects who are not alert or are unresponsive as defined by a score of 2 or 3 on the NIHSS Level of Consciousness question (Question 1a).
* Presence of significant aphasia likely to confound or interfere with completion of the study assessments.
* Presence of a significant pre-existing gait deficit prior to study entry that is likely to confound clinical evaluations
* Presence of pre-existing neurologic or psychiatric disease which is active and not adequately controlled such that it interfered with major activities of daily living immediately prior to the current stroke and is likely to interfere with study participation/visits or confound clinical evaluations.
* The subject poses a significant suicide risk, in the opinion of the investigator.
* Current or chronic history of liver disease, known hepatic or biliary abnormalities (except Gilbert's syndrome or asymptomatic gallstones), or known history of hepatitis B or hepatitis C infection. A positive hepatitis B or hepatitis C result on the GSK labs drawn at baseline/Study Day 1 do not exclude a subject from continuing in the study unless there are associated clinical signs/symptoms of liver disease; however, the subject should be treated as clinically indicated and the GSK Medical Monitor should be contacted for further discussion.
* Presence of either a central or peripheral demyelinating disease, such as multiple sclerosis or IgM monoclonal gammopathy of unknown significance (MGUS).
* Expected death due to the incident stroke, or evidence of a chronic co-morbid condition or unstable acute systemic illness which, in the opinion of the investigator, could shorten the subject's survival such that it would limit his/her ability to complete the study.
* Presence of the following ECG values on baseline ECG: QTc > 500 msec (using either Bazett's formula (QTcB) or Fridericia's formula (QTcF)); or uncorrected QT >600msec (machine or manual over-read). If the ECG indicates a prolonged QTc interval value outside these limits, two further ECGs should be performed during the same sitting and the average QTc value of these triplicate ECGs calculated. If the average value exceeds the stated limits, the subject is not eligible.
* Participation in any investigational rehabilitation paradigm targeting stroke recovery during the duration of this study.
* Have a contraindication to MRI as per local hospital practice/guidelines.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Prior treatment with GSK249320.
* History of sensitivity to Investigational Product excipients (acetate buffer, polysorbate 80 and sodium chloride) that, in the opinion of the investigator or GSK Medical Monitor, contraindicates the subject's participation.
* Pregnant females as determined by positive urine hCG test prior to enrollment.
* Lactating females.
* Subjects considered unwilling or unable to comply with the procedures and study visit schedule outlined in the protocol.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2013-05-18 (Actual); Primary Completion 2014-07-28 (Actual); Study Completion 2014-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (33):
- United States (6):
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Peoria, Illinois
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Nashville, Tennessee
- Canada (5):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Saint-Jérôme, Quebec
- Germany (12):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Friedrichshafen, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Erlangen, Bavaria
  - GSK Investigational Site, Celle, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Osnabrück, Lower Saxony
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Bremen
  - GSK Investigational Site, Hamburg
- United Kingdom (10):
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, Exeter
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, Harrow
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, London
  - GSK Investigational Site, Newcastle upon Tyne
  - GSK Investigational Site, Romford
  - GSK Investigational Site, Salford
  - GSK Investigational Site, Torquay

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Cramer SC, Enney LA, Russell CK, Simeoni M, Thompson TR. Proof-of-Concept Randomized Trial of the Monoclonal Antibody GSK249320 Versus Placebo in Stroke Patients. Stroke. 2017 Mar;48(3):692-698. doi: 10.1161/STROKEAHA.116.014517. Epub 2017 Feb 22. PMID 28228578
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 104615 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104615 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104615 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104615 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104615 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104615 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104615 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 134 participants with Stroke, were randomized to the study. The study was conducted from 18 May 2013 to 28 July 2014 at 30 centers; with 5 in United States, 5 in Canada, 8 in United Kingdom, and 12 in Germany. The ITT population consisted of total 120 participants and the Per Protocol consisted of 104 participants.
Pre-assignment Details: Screening details: This study consisted of a 6 month Core study period and an Extended follow Up period, if required. The study was terminated early at the time of Interim Analysis for reasons of futility. At that time, a total of 134 participants were randomized, of which 133 participants had received at least one dose of study medication.
Groups:
- Placebo: Participants received placebo administered as two intravenous (IV) infusions, the first on Study Day 1 which is 24-72 hours post-stroke onset, and the second on Study Day 6 (+/- 2 days). Each 100 milliliters (mL) IV infusion was delivered over a period of 75 minutes (a 60 minute infusion followed by a 10 to 15 minute flush).
- GSK249320 15 mg/kg: Participants received GSK249320 15 milligrams (mg)/kilogram (kg) administered as two IV infusions, the first on Study Day 1 which is 24-72 post-stroke onset, and the second on Study Day 6 (+/- 2 days). Each 100 mL IV infusion was delivered over a period of 75 minutes (a 60 minute infusion followed by a 10 to 15 minute flush).
Period: Overall Study
Arm/Group | Placebo | GSK249320 15 mg/kg
Started | 68 | 65
Completed | 32 | 32
Not Completed | 36 | 33
Not completed — Physician Decision | 0 | 2
Not completed — Study Closed/Terminated | 25 | 23
Not completed — Adverse event, non-fatal | 2 | 0
Not completed — Consent withdrawn by subject | 6 | 7
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants were administered placebo as two IV infusions, the first on Study Day 1 which was 24-72 hours post-stroke onset, and the second on Study Day 6 (+/- 2 days). Each 100 mL, IV infusion was delivered over a period of 75 minutes (a 60 minute infusion followed by a 10 to 15 minute flush).
- GSK249320 15 mg/kg: Participants received GSK249320 15 mg/kg administered as two IV infusions, the first on Study Day 1 which is 24-72 post-stroke onset, and the second on Study Day 6 (+/- 2 days). Each 100 mL IV infusion was delivered over a period of 75 minutes (a 60 minute infusion followed by a 10 to 15 minute flush).
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK249320 15 mg/kg | Total
Number analyzed (Participants) | 68 | 65 | 133
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (11.2) | 68.2 (11.92) | 67.6 (11.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 31 | 60
  Male | 39 | 34 | 73
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 62 | 62 | 124
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline (BL) to Month 3/ Day 90 in Gait Velocity
Description: Gait is the way or manner in which a person walks. Gait velocity (walking speed) is an objective, quantitative measure of lower extremity motor recovery in individuals who have had a stroke. Participants were asked to walk at their usual pace over a level, indoor 10 meter (m) distance and were allowed to use their normal assistive devices. The time (seconds[s]) taken by the participants to travel the 10 m distance was recorded. Gait velocity (m/s) as assessed by study personnel was derived as: 10 divided by time to walk 10 m. Two trials of gait velocity were conducted at each time point. Change from BL was calculated as the mean Month 3/Day 90 value minus the mean BL value. BL was defined as Day 1. The measure type displayed are posterior means.
Time Frame: BL (Day 1) and Month 3/Day 90
Population: Intent-To-Treat (ITT) population comprised of participants who received at least 1 infusion of investigational product and had at least 1 post-Baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Placebo | GSK249320 15 mg/kg
Number analyzed (Participants) | 60 | 60
m/s | 0.5417 (0.062) | 0.5859 (0.0535)
Statistical Analysis 1: Comparison: Placebo vs GSK249320 15 mg/kg; Credible intervals are displayed as confidence intervals. Posterior means, standard deviations, and credible intervals are provided in the table; Test type: Other; p = 0.713, Bayesian method — P-value presented is the posterior probability that the treatment difference (GSK249320 15mg/kg - placebo) is greater than 0 m/s at Month 3/Day 90; Mean Difference (Net) = 0.0443, 95% CI [-0.119 to 0.2], Standard Error of Mean 0.0809

2. Secondary Outcome: Mean Change From BL to Month 6/ Day 180 in Gait Velocity
Description: Gait is the way or manner in which a person walks. Gait velocity (walking speed) is an objective, quantitative measure of lower extremity motor recovery in individuals who have had a stroke. Participants were asked to walk at their usual pace over a level, indoor 10 m distance and were allowed to use their normal assistive devices. The time (s) taken by the participants to travel the 10 m distance was recorded. Gait velocity (m/s) as assessed by study personnel was derived as: 10 divided by time to walk 10 m. Two trials of gait velocity were conducted at each time point. Change from BL was calculated as the mean Month 3/Day 90 value minus the mean BL value. BL was defined as Day 1. The measure type displayed are posterior means.
Time Frame: BL (Day 1) and Month 6/Day 180
Population: ITT Population.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Placebo | GSK249320 15 mg/kg
Number analyzed (Participants) | 60 | 60
m/s | 0.5442 (0.0665) | 0.6236 (0.0556)
Statistical Analysis 1: Comparison: Placebo vs GSK249320 15 mg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.828, Bayesian method — P-value presented is the posterior probability that the treatment difference (GSK249320 15mg/kg - placebo) is greater than 0 m/s at Month 6/Day 180; Mean Difference (Net) = 0.0794, 95% CI 2-sided [-0.093 to 0.247], Standard Error of Mean 0.0857

3. Secondary Outcome: Number of Participants With Indicated Transition From One Gait Velocity Category to Another Category at the Indicated Time Points
Description: Participants were categorized at each visit into the following gait velocity categories: 0 m/s, >0 to <0.4 m/s, >=0.4 m/s to 0.8 m/s and >0.8m/s. A distinction was made between participants who are too incapacitated to walk (i.e., gait velocity = 0m/s) and participants for whom the gait velocity assessment was not performed due to another reason (i.e., truly missing data). Participants were asked to walk at their usual or normal pace and using their normal assistive devices. Two trials of gait velocity were conducted at each time point. The number of participants transitioning from one gait velocity category to another category was assessed at each post-Baseline visit and was presented in terms of the following transition categories: worsened, no change, improved 1 level, improved 2 levels and improved 3 levels. By-visit sample sizes vary due to missing data or early termination of the study, missing data was not imputed.
Time Frame: BL (Day 1), Month 1/Day 30, Month 2/Day 60, Month 3/Day 90 and Month 6/Day 180.
Population: PP Population consisted of all participants who were included in the ITT population and did not violate protocol with regards to inclusion/exclusion criteria, unblinding, investigational product administration and gait velocity assessments. Only participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo - PP: Participants were administered placebo as two IV infusions, the first on Study Day 1 which was 24-72 hours post-stroke onset, and the second on Study Day 6 (+/- 2 days). Each 100 mL, IV infusion was delivered over a period of 75 minutes (a 60 minute infusion followed by a 10 to 15 minute flush). Placebo - Per Protocol (PP) Population consisted of all participants who were included in the ITT population and did not violate protocol with regards to inclusion/exclusion criteria, unblinding, investigational product administration and gait velocity assessments.
- GSK249320 15 mg/kg - PP: Participants received GSK249320 15 mg/kg administered as two IV infusions, the first on Study Day 1 which is 24-72 post-stroke onset, and the second on Study Day 6 (+/- 2 days). Each 100 mL IV infusion was delivered over a period of 75 minutes (a 60 minute infusion followed by a 10 to 15 minute flush). The GSK249320 15 mg/kg - PP Population consisted of all participants who were included in the ITT population and did not violate protocol with regards to inclusion/exclusion criteria, unblinding, investigational product administration and gait velocity assessments.
Arm/Group | Placebo - PP | GSK249320 15 mg/kg - PP
Number analyzed (Participants) | 52 | 52
Participants
  Day 30, Worsened: number analyzed (Participants) | 48 | 49
  Day 30, Worsened | 1 | 0
  Day 30, No Change: number analyzed (Participants) | 48 | 49
  Day 30, No Change | 19 | 18
  Day 30, Improved 1 Levels: number analyzed (Participants) | 48 | 49
  Day 30, Improved 1 Levels | 11 | 11
  Day 30, Improved 2 Levels: number analyzed (Participants) | 48 | 49
  Day 30, Improved 2 Levels | 9 | 9
  Day 30, Improved 3 Levels: number analyzed (Participants) | 48 | 49
  Day 30, Improved 3 Levels | 8 | 11
  Day 60, Worsened: number analyzed (Participants) | 42 | 42
  Day 60, Worsened | 0 | 0
  Day 60, No Change: number analyzed (Participants) | 42 | 42
  Day 60, No Change | 13 | 14
  Day 60, Improved 1 Level: number analyzed (Participants) | 42 | 42
  Day 60, Improved 1 Level | 14 | 11
  Day 60, Improved 2 Levels: number analyzed (Participants) | 42 | 42
  Day 60, Improved 2 Levels | 6 | 7
  Day 60, Improved 3 Levels: number analyzed (Participants) | 42 | 42
  Day 60, Improved 3 Levels | 9 | 10
  Day 90, Worsened: number analyzed (Participants) | 42 | 41
  Day 90, Worsened | 1 | 0
  Day 90, No Change: number analyzed (Participants) | 42 | 41
  Day 90, No Change | 9 | 8
  Day 90, Improved 1 Level: number analyzed (Participants) | 42 | 41
  Day 90, Improved 1 Level | 12 | 14
  Day 90, Improved 2 Levels: number analyzed (Participants) | 42 | 41
  Day 90, Improved 2 Levels | 10 | 7
  Day 90, Improved 3 Levels: number analyzed (Participants) | 42 | 41
  Day 90, Improved 3 Levels | 10 | 12
  Day 180, Worsened: number analyzed (Participants) | 36 | 39
  Day 180, Worsened | 1 | 0
  Day 180, No Change: number analyzed (Participants) | 36 | 39
  Day 180, No Change | 7 | 6
  Day 180, Improved 1 Level: number analyzed (Participants) | 36 | 39
  Day 180, Improved 1 Level | 9 | 14
  Day 180, Improved 2 Levels: number analyzed (Participants) | 36 | 39
  Day 180, Improved 2 Levels | 11 | 5
  Day 180, Improved 3 Levels: number analyzed (Participants) | 36 | 39
  Day 180, Improved 3 Levels | 8 | 14

4. Secondary Outcome: Change From BL in Dexterity as Measured by Box and Blocks Test
Description: Dexterity is ability of person to use hands skillfully in performing a task. Box and Blocks test is an objective, gross manual dexterity test in individuals with upper limb impairments. Participants were asked to move small wooden blocks from one side of a partitioned box to other. The score was determined by number of blocks transferred within a 60 second time period. Both affected and unaffected arms were tested, starting with the unaffected arm. Change from BL was calculated as the individual post- BL value minus BL value. A higher number of displaced blocks indicated a better gross dexterity and a low number of displaced blocks indicated poor gross dexterity. It was analyzed using fixed effects for treatment, visit, treatment by visit interaction, sex, age, Baseline National Institute of Health stroke scale (NIHSS) total score, BL number of blocks transferred by the affected and unaffected arms, country and presence of concomitant medications that potentially impact recovery.
Time Frame: BL (Day 1), Month 1/Day 30, Month 2/Day 60, Month 3/Day 90 and Month 6/Day 180
Population: PP Population.
Measure: Least Squares Mean (Standard Error); unit: Number of blocks
Groups:
- Placebo - PP: Participants were administered placebo as two IV infusions, the first on Study Day 1 which was 24-72 hours post-stroke onset, and the second on Study Day 6 (+/- 2 days). Each 100 mL, IV infusion was delivered over a period of 75 minutes (a 60 minute infusion followed by a 10 to 15 minute flush). Placebo PP Population consisted of all participants who were included in the ITT population and did not violate protocol with regards to inclusion/exclusion criteria, unblinding, investigational product administration and gait velocity assessments.
Arm/Group | Placebo - PP | GSK249320 15 mg/kg - PP
Number analyzed (Participants) | 52 | 52
Number of blocks
  Day 30 | 10.130 (2.195) | 12.538 (1.587)
  Day 60 | 11.469 (2.345) | 14.484 (1.6)
  Day 90 | 15.196 (2.962) | 17.631 (1.926)
  Day 180 | 14.869 (2.839) | 18.813 (2.11)
Statistical Analysis 1: Comparison: Placebo - PP vs GSK249320 15 mg/kg - PP; Statistical data for Day 30. The point estimate and confidence interval are for the adjusted mean difference based on least square estimates; Test type: Other; Mean Difference (Net) = 2.408, 95% CI 2-sided [-3.067 to 7.883], Standard Error of Mean 2.7495
Statistical Analysis 2: Comparison: Placebo - PP vs GSK249320 15 mg/kg - PP; Statistical data for Day 60. The point estimate and confidence interval are for the adjusted mean difference based on least square estimates; Test type: Other; Mean Difference (Net) = 3.015, 95% CI 2-sided [-2.704 to 8.735], Standard Error of Mean 2.8732
Statistical Analysis 3: Comparison: Placebo - PP vs GSK249320 15 mg/kg - PP; Statistical data for Day 90. The point estimate and confidence interval are for the adjusted mean difference based on least square estimates; Test type: Other; Mean Difference (Net) = 2.435, 95% CI 2-sided [-4.668 to 9.538], Standard Error of Mean 3.5633
Statistical Analysis 4: Comparison: Placebo - PP vs GSK249320 15 mg/kg - PP; Statistical data for Day 180. The point estimate and confidence interval are for the adjusted mean difference based on least square estimates; Test type: Other; Mean Difference (Net) = 3.944, 95% CI 2-sided [-3.15 to 11.037], Standard Error of Mean 3.5635

5. Secondary Outcome: Number of Participants Experiencing Falls
Description: The number of participants who experienced at least one fall between BL to Day 90 and BL to Day 180 is summarized.
Time Frame: BL (Day 1) Day 90 and Day 180
Population: Safety population is defined as participants who had received at least one infusion of investigational product.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo - Safety: Participants received placebo administered as two IV infusions, the first on Study Day 1 which is 24-72 hours post-stroke onset, and the second on Study Day 6 (+/- 2 days). Each 100 mL IV infusion was delivered over a period of 75 minutes (a 60 minute infusion followed by a 10 to 15 minute flush). The Safety Population included all participants who received at least one infusion of investigational product.
- GSK249320 15 mg/kg - Safety: Participants received GSK249320 15 mg/kg administered as two IV infusions, the first on Study Day 1 which is 24-72 post-stroke onset, and the second on Study Day 6 (+/- 2 days). Each 100 mL IV infusion was delivered over a period of 75 minutes (a 60 minute infusion followed by a 10 to 15 minute flush). The Safety Population included all participants who received at least one infusion of investigational product.
Arm/Group | Placebo - Safety | GSK249320 15 mg/kg - Safety
Number analyzed (Participants) | 68 | 65
Participants
  Baseline to Day 90 | 15 | 12
  Baseline to Day 180 | 18 | 16

6. Secondary Outcome: Number of Falls Over Time
Description: The number of participants who experienced 1, 2, 3 or >=4 falls between BL to Day 90 and BL to Day 180 is summarized. By-visit sample sizes vary due to missing data or early termination of the study. The participants who experienced atleast one-fall were reported
Time Frame: BL (Day 1), Day 90 and Day 180
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo - Safety | GSK249320 15 mg/kg - Safety
Number analyzed (Participants) | 68 | 65
Participants
  Baseline to Day 90, 1 Fall | 8 | 6
  Baseline to Day 90, 2 Falls | 3 | 3
  Baseline to Day 90, 3 Falls | 0 | 2
  Baseline to Day 90, >=4 Falls | 4 | 1
  Baseline to Day 180, 1 Fall | 7 | 9
  Baseline to Day 180, 2 Falls | 6 | 2
  Baseline to Day 180, 3 Falls | 1 | 2
  Baseline to Day 180, >=4 Falls | 4 | 3

7. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A SAE is any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect or all events of possible drug-induced liver injury with hyperbilirubinaemia. Medical or scientific judgment is exercised in other situations.
Time Frame: Up to 14 months
Population: Safety population.
Measure: Count of Participants; unit: Participants
Groups:
- GSK249320 15/mg: Participants received GSK249320 15 mg/kg administered as two IV infusions, the first on Study Day 1 which is 24-72 post-stroke onset, and the second on Study Day 6 (+/- 2 days). Each 100 mL IV infusion was delivered over a period of 75 minutes (a 60 minute infusion followed by a 10 to 15 minute flush).
Arm/Group | Placebo | GSK249320 15/mg
Number analyzed (Participants) | 68 | 65
Participants
  Any AE | 57 | 49
  Any SAE | 16 | 9

8. Secondary Outcome: Number of Participants With Events Common to Stroke
Description: Events common to stroke were those events that commonly occurred after a stroke and are generally associated with the underlying stroke or the progression of stroke. These included joint or soft tissue pain, bladder incontinence, depression/mood disorder, urinary tract infection, dysphagia, bowel incontinence, dysarthia, confusion, spasticity, limb edema, aspiration pneumonia, hemorrhagic transformation (symptomatic or asymptomatic), pressure ulcers, progression of stroke, malnutrition, deep vein thrombosis, brain herniation, pulmonary embolism, seizures, and falls.
Time Frame: From Day 1 until early withdrawal, death, Month 6/Day 180
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK249320 15/mg
Number analyzed (Participants) | 68 | 65
Participants
  Joint or soft tissue pain | 19 | 22
  Bladder Incontinence | 11 | 23
  Depression/Mood Disorder | 17 | 16
  Urinary tract infection | 17 | 13
  Dysphagia | 12 | 12
  Bowel Incontinence | 11 | 12
  Dysarthia | 11 | 11
  Confusion | 8 | 13
  Spasticity | 9 | 9
  Limb edema | 5 | 12
  Aspiration Pneumonia | 5 | 3
  Hemorrhagic Transformation | 4 | 4
  Pressure Ulcers | 3 | 2
  Progression of Stroke | 2 | 2
  Malnutrition | 1 | 2
  Deep vein thrombosis | 2 | 0
  Brain Herniation | 0 | 1
  Pulmonary embolism | 1 | 0
  Seizures | 0 | 1
  Falls | 18 | 16

9. Secondary Outcome: Change From BL in Vital Signs- Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Safety was measured by monitoring vital signs including blood pressure. The BL for DBP and SBP was the value of pre-dose assessment on Day 1. Change from BL was calculated as the individual post-Baseline value minus the BL value. By-visit sample sizes vary due to missing data or early termination of the study.
Time Frame: BL (Day 1) , Day 6, Day 180 and early withdrawal (EW) visit
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Placebo - Safety | GSK249320 15 mg/kg - Safety
Number analyzed (Participants) | 68 | 65
Millimeters of mercury
  DBP, Day 1 Post-dose | 1.7 (10.58) | 0.5 (10.14)
  DBP, Day 6 Pre-dose: number analyzed (Participants) | 60 | 59
  DBP, Day 6 Pre-dose | 0.2 (16.52) | -1.1 (11.98)
  DBP, Day 6 Post-dose: number analyzed (Participants) | 58 | 57
  DBP, Day 6 Post-dose | 2.4 (15.06) | 1.9 (16.36)
  DBP, Day 180: number analyzed (Participants) | 27 | 28
  DBP, Day 180 | 8.1 (13.97) | 5.0 (14.60)
  DBP, EW visit: number analyzed (Participants) | 24 | 22
  DBP, EW visit | -5.0 (15.55) | 1.8 (15.05)
  SBP, Day 1 Post-dose | 3.1 (16.15) | 0.7 (11.81)
  SBP, Day 6 Pre-dose: number analyzed (Participants) | 60 | 59
  SBP, Day 6 Pre-dose | -3.5 (26.46) | -6.0 (20.13)
  SBP, Day 6 Post-dose: number analyzed (Participants) | 58 | 57
  SBP, Day 6 Post-dose | -0.9 (24.59) | -2.0 (20.14)
  SBP, Day 180: number analyzed (Participants) | 27 | 28
  SBP, Day 180 | -6.4 (22.96) | -6.4 (27.79)
  SBP, EW visit: number analyzed (Participants) | 24 | 22
  SBP, EW visit | -15.2 (29.08) | -0.0 (25.42)

10. Secondary Outcome: Change From BL in Vitals Signs-Heart Rate
Description: Safety was measured by monitoring vital signs including heart rate. The BL for heart rate was the value of pre-dose assessment on Day 1. Change from BL was calculated as the individual post-BL value minus the BL value. By-visit sample sizes vary due to missing data or early termination of the study. BL was defined as Day 1.
Time Frame: Day 1, Day 6, Day 180 and EW visit
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo - Safety | GSK249320 15 mg/kg - Safety
Number analyzed (Participants) | 68 | 65
Beats per minute
  Day 1 Post-dose: number analyzed (Participants) | 67 | 65
  Day 1 Post-dose | 0.9 (8.68) | 0.7 (7.98)
  Day 6 Pre-dose: number analyzed (Participants) | 60 | 59
  Day 6 Pre-dose | -1.8 (13.03) | -0.4 (17.47)
  Day 6 Post-dose: number analyzed (Participants) | 58 | 57
  Day 6 Post-dose | -3.9 (12.09) | -3.1 (15.30)
  Day 180: number analyzed (Participants) | 27 | 28
  Day 180 | -0.3 (17.50) | -3.0 (15.48)
  EW visit: number analyzed (Participants) | 24 | 22
  EW visit | 3.3 (15.47) | -2.1 (15.40)

11. Secondary Outcome: Change From BL in ECG Parameter-Heart Rate
Description: A single 12-lead ECG was obtained at each time point that measured heart rate. BL was the value obtained on Day 1. Change from BL was calculated as the individual post-Baseline value minus the BL value. By-visit sample sizes vary due to missing data or early termination of the study.
Time Frame: BL (Day 1) Day 6, Day 30 and EW visit
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo - Safety | GSK249320 15 mg/kg - Safety
Number analyzed (Participants) | 68 | 65
Beats per minute
  Day 6, n=60, 58: number analyzed (Participants) | 60 | 58
  Day 6, n=60, 58 | -3.4 (17.57) | -4.9 (15.37)
  Day 30, n=46, 50: number analyzed (Participants) | 46 | 50
  Day 30, n=46, 50 | -3.4 (19.81) | 0.9 (16)
  EW Visit, n=16, 16: number analyzed (Participants) | 16 | 16
  EW Visit, n=16, 16 | -5.4 (16.82) | -10.3 (29.58)

12. Secondary Outcome: Change From BL in ECG Parameters
Description: A single 12-lead ECG was obtained at each time point and the following ECG intervals were determined: PR, QRS, QT, RR and corrected QT (QTc), QT interval corrected by Bazett's formula (QTcB), QT interval corrected by Fridericia's formula (QTcF). BL for ECG parameters was the value of Day 1. Change from BL was calculated as the individual post-Baseline value minus the BL value. By-visit sample sizes vary due to missing data or early termination of the study.
Time Frame: BL (Day 1), Day 6, Day 30 and EW visit
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Placebo - Safety | GSK249320 15 mg/kg - Safety
Number analyzed (Participants) | 68 | 65
Milliseconds
  PR, Day 6: number analyzed (Participants) | 50 | 46
  PR, Day 6 | -1.0 (30.47) | -0.8 (20.02)
  PR, Day 30: number analyzed (Participants) | 38 | 40
  PR, Day 30 | -5.9 (36.05) | -3.5 (42.08)
  PR, EW Visit: number analyzed (Participants) | 10 | 14
  PR, EW Visit | -0.4 (21.01) | 3.1 (33.96)
  QRS, Day 6: number analyzed (Participants) | 60 | 57
  QRS, Day 6 | 4.9 (15.75) | -4.0 (44.11)
  QRS, Day 30: number analyzed (Participants) | 46 | 50
  QRS, Day 30 | 3.4 (10.97) | 1.1 (17.74)
  QRS, EW Visit: number analyzed (Participants) | 16 | 16
  QRS, EW Visit | 2.6 (27.47) | -23.7 (81.24)
  RR, Day 6: number analyzed (Participants) | 53 | 53
  RR, Day 6 | 61.1 (246.84) | 12.9 (154.09)
  RR, Day 30: number analyzed (Participants) | 40 | 45
  RR, Day 30 | 80.5 (245.31) | -21.8 (181.99)
  RR, EW Visit: number analyzed (Participants) | 13 | 16
  RR, EW Visit | -21.6 (164.19) | 85.6 (349.82)
  QT, Day 6: number analyzed (Participants) | 60 | 57
  QT, Day 6 | 10.4 (40.86) | 9.4 (36.46)
  QT, Day 30: number analyzed (Participants) | 46 | 49
  QT, Day 30 | 4.1 (43.59) | -12.1 (42.06)
  QT, EW Visit: number analyzed (Participants) | 16 | 15
  QT, EW Visit | 20.8 (37.16) | 43.7 (93.85)
  QTc, Day 6: number analyzed (Participants) | 58 | 58
  QTc, Day 6 | 2.9 (30.70) | 6.8 (43.87)
  QTc, Day 30: number analyzed (Participants) | 45 | 50
  QTc, Day 30 | -1.3 (32.92) | -2.2 (39.49)
  QTc, EW Visit: number analyzed (Participants) | 16 | 16
  QTc, EW Visit | 7.1 (27.75) | 8.9 (69.58)
  QTcB, Day 6: number analyzed (Participants) | 53 | 51
  QTcB, Day 6 | 2.2 (124.73) | 4.5 (46.49)
  QTcB, Day 30: number analyzed (Participants) | 40 | 44
  QTcB, Day 30 | -31.9 (120.26) | -13.9 (79.33)
  QTcB, EW Visit: number analyzed (Participants) | 13 | 14
  QTcB, EW Visit | 28.2 (37.06) | 6.9 (52.02)
  QTcF, Day 6: number analyzed (Participants) | 53 | 51
  QTcF, Day 6 | 4.3 (74.12) | 5.7 (33.25)
  QTcF, Day 30: number analyzed (Participants) | 40 | 44
  QTcF, Day 30 | -16.9 (75.41) | -12.0 (58.16)
  QTcF, EW Visit: number analyzed (Participants) | 13 | 14
  QTcF, EW Visit | 26.0 (31.85) | 18.3 (62.78)

13. Secondary Outcome: Change From BL in Clinical Chemistry- Albumin and Total Protein
Description: ALB and TP were measured at BL, Day 6, Day 30, Day 90 and Day 180. Baseline was the value obtained on Day 1. Change from BL was calculated as the individual post-Baseline value minus the BL value. By-visit sample sizes vary due to missing data or early termination of the study.
Time Frame: BL (Day 1), Day 6, Day 30, Day 90 and Day 180
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Placebo - Safety | GSK249320 15 mg/kg - Safety
Number analyzed (Participants) | 68 | 65
Grams per liter
  ALB, Day 6: number analyzed (Participants) | 56 | 57
  ALB, Day 6 | 0.0 (3.02) | -0.2 (3.67)
  ALB, Day 30: number analyzed (Participants) | 44 | 47
  ALB, Day 30 | 1.0 (3.44) | 3.0 (5.50)
  ALB, Day 90: number analyzed (Participants) | 32 | 38
  ALB, Day 90 | 2.3 (3.23) | 4.4 (5.14)
  ALB, Day 180: number analyzed (Participants) | 23 | 24
  ALB, Day 180 | 2.3 (3.80) | 5.3 (3.86)
  TP, Day 6: number analyzed (Participants) | 56 | 57
  TP, Day 6 | 1.0 (4.64) | 0.9 (5.90)
  TP, Day 30: number analyzed (Participants) | 44 | 47
  TP, Day 30 | 2.7 (5.13) | 5.6 (8.11)
  TP, Day 90: number analyzed (Participants) | 32 | 38
  TP, Day 90 | 3.1 (4.92) | 6.5 (7.34)
  TP, Day 180: number analyzed (Participants) | 23 | 24
  TP, Day 180 | 4.4 (5.07) | 7.6 (5.89)

14. Secondary Outcome: Change From BL in Clinical Chemistry-urea/Blood Urea Nitrogen (BUN), Sodium (Na), Potassium (K), Glucose (Gluc), Chloride (Cl), Calcium (Ca)
Description: Ca, Cl, Gluc, K, Na and BUN were measured at BL, Day 6, Day 30, Day 90 and Day 180. BL was the value obtained on Day 1. Change from BL was calculated as the individual post-Baseline value minus the BL value. By-visit sample sizes vary due to missing data or early termination of the study.
Time Frame: BL (Day 1), Day 6, Day 30, Day 90 and Day 180
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Placebo - Safety | GSK249320 15 mg/kg - Safety
Number analyzed (Participants) | 68 | 65
Millimoles per liter
  Ca, Day 6: number analyzed (Participants) | 56 | 54
  Ca, Day 6 | 0.042 (0.1163) | 0.059 (0.1564)
  Ca, Day 30: number analyzed (Participants) | 44 | 46
  Ca, Day 30 | 0.091 (0.1254) | 0.158 (0.1985)
  Ca, Day 90: number analyzed (Participants) | 32 | 37
  Ca, Day 90 | 0.093 (0.1092) | 0.186 (0.1960)
  Ca, Day 180: number analyzed (Participants) | 23 | 23
  Ca, Day 180 | 0.087 (0.1053) | 0.182 (0.1315)
  Cl, Day 6: number analyzed (Participants) | 56 | 57
  Cl, Day 6 | -0.9 (3.13) | -1.4 (4.08)
  Cl, Day 30: number analyzed (Participants) | 44 | 47
  Cl, Day 30 | -1.6 (3.72) | -3.1 (5.01)
  Cl, Day 90: number analyzed (Participants) | 32 | 38
  Cl, Day 90 | -1.3 (3.02) | -2.7 (4.67)
  Cl, Day 180: number analyzed (Participants) | 23 | 24
  Cl, Day 180 | -1.4 (2.48) | -3.4 (3.93)
  Gluc, Day 6: number analyzed (Participants) | 56 | 57
  Gluc, Day 6 | 0.21 (3.123) | -0.35 (2.619)
  Gluc, Day 30: number analyzed (Participants) | 44 | 47
  Gluc, Day 30 | -0.93 (2.611) | -0.45 (2.476)
  Gluc, Day 90: number analyzed (Participants) | 32 | 38
  Gluc, Day 90 | -1.12 (2.075) | -0.38 (2.170)
  Gluc, Day 180: number analyzed (Participants) | 23 | 24
  Gluc, Day 180 | -1.09 (3.045) | -1.02 (2.136)
  K, Day 6: number analyzed (Participants) | 55 | 54
  K, Day 6 | 0.17 (0.384) | 0.21 (0.452)
  K, Day 30: number analyzed (Participants) | 43 | 46
  K, Day 30 | 0.37 (0.487) | 0.30 (0.429)
  K, Day 90: number analyzed (Participants) | 31 | 37
  K, Day 90 | 0.36 (0.477) | 0.39 (0.404)
  K, Day 180: number analyzed (Participants) | 22 | 23
  K, Day 180 | 0.33 (0.517) | 0.54 (0.472)
  Na, Day 6: number analyzed (Participants) | 56 | 57
  Na, Day 6 | 0.1 (2.82) | 0.0 (2.83)
  Na, Day 30: number analyzed (Participants) | 44 | 47
  Na, Day 30 | -0.3 (2.64) | -0.8 (3.21)
  Na, Day 90: number analyzed (Participants) | 32 | 38
  Na, Day 90 | 0.4 (1.87) | -0.7 (2.91)
  Na, Day 180: number analyzed (Participants) | 23 | 24
  Na, Day 180 | 0.5 (2.04) | -1.2 (2.90)
  Urea/BUN, Day 6: number analyzed (Participants) | 56 | 57
  Urea/BUN, Day 6 | 1.57 (2.392) | 1.61 (2.541)
  Urea/BUN, Day 30: number analyzed (Participants) | 44 | 47
  Urea/BUN, Day 30 | 1.09 (2.673) | 2.19 (5.436)
  Urea/BUN, Day 90: number analyzed (Participants) | 32 | 38
  Urea/BUN, Day 90 | 1.02 (2.310) | 1.04 (2.655)
  Urea/BUN, Day 180: number analyzed (Participants) | 23 | 24
  Urea/BUN, Day 180 | 0.51 (2.364) | 1.04 (3.502)

15. Secondary Outcome: Change From BL in Alkaline Phosphatase (ALP), Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST)
Description: ALP, ALT and AST were measured at BL, Day 6, Day 30, Day 90 and Day 180. BL was the value obtained on Day 1. Change from BL was calculated as the individual post-Baseline value minus the BL value. By-visit sample sizes vary due to missing data or early termination of the study.
Time Frame: BL (Day 1), Day 6, Day 30, Day 90 and Day 180
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Placebo - Safety | GSK249320 15 mg/kg - Safety
Number analyzed (Participants) | 68 | 65
International units per liter
  ALP, Day 6: number analyzed (Participants) | 56 | 57
  ALP, Day 6 | 7.7 (20.05) | 6.2 (16.4)
  ALP, Day 30: number analyzed (Participants) | 44 | 47
  ALP, Day 30 | 11.7 (21.47) | 19.5 (35.87)
  ALP, Day 90: number analyzed (Participants) | 32 | 38
  ALP, Day 90 | 8.6 (27.18) | 6.7 (18.01)
  ALP, Day 180: number analyzed (Participants) | 23 | 24
  ALP, Day 180 | 8.9 (12.73) | 4.0 (17.63)
  ALT, Day 6: number analyzed (Participants) | 56 | 57
  ALT, Day 6 | 11.4 (25.92) | 10.7 (16.22)
  ALT, Day 30: number analyzed (Participants) | 44 | 47
  ALT, Day 30 | 7.9 (19.02) | 10.6 (27.84)
  ALT, Day 90: number analyzed (Participants) | 32 | 38
  ALT, Day 90 | -0.8 (16.14) | 3.2 (11.21)
  ALT, Day 180: number analyzed (Participants) | 23 | 24
  ALT, Day 180 | -2.0 (12.83) | 1.4 (10.66)
  AST, Day 6: number analyzed (Participants) | 56 | 54
  AST, Day 6 | 7.9 (26.39) | 2.5 (15.52)
  AST, Day 30: number analyzed (Participants) | 44 | 46
  AST, Day 30 | 0.2 (14.24) | -0.9 (13.18)
  AST, Day 90: number analyzed (Participants) | 32 | 37
  AST, Day 90 | -6.1 (11.78) | -5.2 (13.33)
  AST, Day 180: number analyzed (Participants) | 23 | 23
  AST, Day 180 | -3.2 (7.13) | -5.0 (9.70)

16. Secondary Outcome: Change From BL in Clinical Chemistry- Direct Bilirubin, Total Bilirubin, Creatinine
Description: Direct bilirubin, total bilirubin and creatinine were measured at BL, Day 6, Day 30, Day 90 and Day 180. BL was the value obtained on Day 1. Change from BL was calculated as the individual post-Baseline value minus the BL value. By-visit sample sizes vary due to missing data or early termination of the study.
Time Frame: BL (Day 1), Day 6, Day 30, Day 90 and Day 180
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Placebo - Safety | GSK249320 15 mg/kg - Safety
Number analyzed (Participants) | 68 | 65
Micromoles per liter
  direct bilirubin, Day 6: number analyzed (Participants) | 56 | 57
  direct bilirubin, Day 6 | 0.3 (3.81) | -0.0 (1.58)
  direct bilirubin, Day 30: number analyzed (Participants) | 44 | 47
  direct bilirubin, Day 30 | -1.0 (1.93) | -0.4 (1.48)
  direct bilirubin, Day 90: number analyzed (Participants) | 32 | 38
  direct bilirubin, Day 90 | -1.5 (1.92) | -0.5 (1.62)
  direct bilirubin, Day 180: number analyzed (Participants) | 23 | 24
  direct bilirubin, Day 180 | -1.2 (1.59) | -0.1 (1.38)
  total bilirubin, Day 6: number analyzed (Participants) | 56 | 57
  total bilirubin, Day 6 | -1.5 (3.76) | -1.8 (5.90)
  total bilirubin, Day 30: number analyzed (Participants) | 44 | 47
  total bilirubin, Day 30 | -4.6 (4.90) | -3.0 (4.85)
  total bilirubin, Day 90: number analyzed (Participants) | 32 | 38
  total bilirubin, Day 90 | -4.9 (4.75) | -3.5 (5.59)
  total bilirubin, Day 180: number analyzed (Participants) | 23 | 24
  total bilirubin, Day 180 | -4.6 (4.83) | -3.8 (5.28)
  creatinine, Day 6: number analyzed (Participants) | 56 | 57
  creatinine, Day 6 | 2.35 (20.520) | 3.48 (16.778)
  creatinine, Day 30: number analyzed (Participants) | 44 | 47
  creatinine, Day 30 | 4.94 (31.767) | 9.79 (28.329)
  creatinine, Day 90: number analyzed (Participants) | 32 | 38
  creatinine, Day 90 | 6.69 (18.980) | 3.09 (15.387)
  creatinine, Day 180: number analyzed (Participants) | 23 | 24
  creatinine, Day 180 | 5.07 (12.925) | 0.24 (13.857)

17. Secondary Outcome: Change From BL in Eosinophils (EOS), Lymphocytes (LYM), Total Absolute Neutrophil Count (ANC), Platelet (PLT) Count, White Blood Cell (WBC) Count
Description: EOS, LYM, Total ANC, PLT count and WBC count were measured at BL, Day 6, Day 30, Day 90 and Day 180. BL was the value obtained on Day 1. Change from BL was calculated as the individual post-Baseline value minus the BL value.By-visit sample sizes vary due to missing data or early termination of the study.
Time Frame: BL (Day 1), Day 6, Day 30, Day 90 and Day 180
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Giga (10^9 cells) per liter
Arm/Group | Placebo - Safety | GSK249320 15 mg/kg - Safety
Number analyzed (Participants) | 68 | 65
Giga (10^9 cells) per liter
  EOS, Day 6: number analyzed (Participants) | 48 | 51
  EOS, Day 6 | 0.049 (0.1153) | 0.082 (0.1692)
  EOS, Day 30: number analyzed (Participants) | 38 | 44
  EOS, Day 30 | 0.058 (0.2207) | 0.086 (0.1318)
  EOS, Day 90: number analyzed (Participants) | 28 | 35
  EOS, Day 90 | 0.058 (0.1175) | 0.058 (0.1149)
  EOS, Day 180: number analyzed (Participants) | 20 | 22
  EOS, Day 180 | 0.045 (0.1314) | 0.048 (0.1206)
  LYM, Day 6: number analyzed (Participants) | 48 | 51
  LYM, Day 6 | -0.046 (0.3904) | -0.030 (0.6750)
  LYM, Day 30: number analyzed (Participants) | 38 | 44
  LYM, Day 30 | 0.026 (0.4666) | -0.002 (0.5728)
  LYM, Day 90: number analyzed (Participants) | 28 | 35
  LYM, Day 90 | 0.066 (0.4110) | 0.236 (0.5854)
  LYM, Day 180: number analyzed (Participants) | 20 | 22
  LYM, Day 180 | 0.017 (0.5005) | 0.075 (0.5919)
  Total ANC, Day 6: number analyzed (Participants) | 48 | 51
  Total ANC, Day 6 | -0.375 (2.2795) | -0.756 (2.5842)
  Total ANC, Day 30: number analyzed (Participants) | 38 | 44
  Total ANC, Day 30 | -1.486 (2.4578) | -0.581 (4.7282)
  Total ANC, Day 90: number analyzed (Participants) | 28 | 35
  Total ANC, Day 90 | -1.469 (2.1498) | -1.455 (2.3515)
  Total ANC, Day 180: number analyzed (Participants) | 20 | 22
  Total ANC, Day 180 | -2.202 (2.7396) | -0.579 (1.6956)
  PLT Count, Day 6: number analyzed (Participants) | 47 | 48
  PLT Count, Day 6 | 17.4 (37.57) | 32.4 (41.01)
  PLT Count, Day 30: number analyzed (Participants) | 37 | 42
  PLT Count, Day 30 | 40.5 (62.89) | 47.6 (44.23)
  PLT Count, Day 90: number analyzed (Participants) | 28 | 34
  PLT Count, Day 90 | 33.2 (53.36) | 60.4 (56.30)
  PLT Count, Day 180: number analyzed (Participants) | 20 | 22
  PLT Count, Day 180 | 19.9 (35.91) | 35.9 (39.15)
  WBC Count,Day 6: number analyzed (Participants) | 48 | 51
  WBC Count,Day 6 | -0.40 (2.294) | -0.78 (2.288)
  WBC Count, Day 30: number analyzed (Participants) | 38 | 44
  WBC Count, Day 30 | -1.46 (2.524) | -0.54 (4.819)
  WBC Count, Day 90: number analyzed (Participants) | 28 | 35
  WBC Count, Day 90 | -1.45 (2.017) | -1.28 (2.119)
  WBC Count, Day 180: number analyzed (Participants) | 20 | 22
  WBC Count, Day 180 | -2.15 (2.496) | -0.55 (1.943)

18. Secondary Outcome: Change From BL in Hematology- Hemoglobin
Description: Hemoglobin was measured at BL Day 6, Day 30, Day 90 and Day 180. BL was the value obtained on Day 1. Change from BL was calculated as the individual post-Baseline value minus the BL value. . By-visit sample sizes vary due to missing data or early termination of the study.
Time Frame: BL (Day 1), Day 6, Day 30, Day 90 and Day 180
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Placebo - Safety | GSK249320 15 mg/kg - Safety
Number analyzed (Participants) | 68 | 65
Grams per liter
  Day 6: number analyzed (Participants) | 48 | 51
  Day 6 | -0.1 (9.55) | 2.4 (10.21)
  Day 30: number analyzed (Participants) | 38 | 44
  Day 30 | -1.0 (13.19) | 3.8 (14.84)
  Day 90: number analyzed (Participants) | 28 | 35
  Day 90 | -4.1 (16.61) | 4.7 (15.91)
  Day 180: number analyzed (Participants) | 20 | 22
  Day 180 | -6.2 (17.70) | 7.6 (13.45)

19. Secondary Outcome: Change From Baseline in Hematology- Hematocrit
Description: Hematocrit was measured at Baseline, Day 6, Day 30, Day 90 and Day 180. BL was the value obtained on Day 1. Change from BL was calculated as the individual post-Baseline value minus the BL value.By-visit sample sizes vary due to missing data or early termination of the study.
Time Frame: BL (Day 1), Day 6, Day 30, Day 90 and Day 180
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo - Safety | GSK249320 15 mg/kg - Safety
Number analyzed (Participants) | 68 | 65
Ratio
  Day 6: number analyzed (Participants) | 48 | 51
  Day 6 | 0.00096 (0.032094) | 0.00896 (0.032858)
  Day 30: number analyzed (Participants) | 38 | 44
  Day 30 | -0.00350 (0.040669) | 0.01116 (0.046146)
  Day 90: number analyzed (Participants) | 28 | 35
  Day 90 | -0.01446 (0.053418) | 0.01329 (0.049054)
  Day 180: number analyzed (Participants) | 20 | 22
  Day 180 | -0.02455 (0.056181) | 0.01909 (0.043139)

20. Secondary Outcome: Change From BL in NIHSS Total Score
Description: The NIHSS is a 15 item, standardized, disease-specific, deficit scale which measures neurological impairment (level of consciousness, eye movements, visual fields, facial symmetry, motor strength (arm and leg), coordination, sensation, language (aphasia and dysarthria), and neglect) and is used to quantify participant status by measuring the severity of the stroke as assessed by NIHSS certified study personnel. The total NIHSS score is calculated as the sum of responses to the 15 items. The total NIHSS score ranges from 0-42, with a higher score indicative of a more severe impairment. By-visit sample sizes vary due to missing data or early termination of the study. Change from BL was calculated as the individual post-Baseline value minus the BL value. BL was defined as the value at Day 1.
Time Frame: BL (Day 1), Day 30, Day 90 and Day 180
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo - Safety | GSK249320 15 mg/kg - Safety
Number analyzed (Participants) | 68 | 65
Scores on a scale
  Day 1 | 10.0 (4.40) | 9.8 (3.79)
  Day 30: number analyzed (Participants) | 52 | 55
  Day 30 | 6.4 (4.40) | 5.7 (4.66)
  Day 90: number analyzed (Participants) | 40 | 45
  Day 90 | 5.0 (3.83) | 4.8 (4.89)
  Day 180: number analyzed (Participants) | 27 | 30
  Day 180 | 3.9 (3.22) | 4.2 (3.87)

21. Secondary Outcome: Number of Participants With Suicidal Ideation Via Columbia Suicide Severity Rating Scale (CSSRS)
Description: C-SSRS is a clinician-rated scale that evaluates severity and change of suicidality by integrating both suicidality behavior and ideation. For Suicidal Ideation (SI), participants were scored non-suicidal:0, wish to be dead:1, non-specific active suicidal thoughts:2, active suicidal ideation with associated thoughts of methods without intent:3, active suicidal ideation with some intent to act on suicidal thoughts without clear plan:4, active suicidal ideation with plan and intent:5 (most severe). SI intensity total score was the sum of suicidal ideation severity rating scores for frequency, duration, controllability, deterrents, and reasons for ideation. For each item, each participant got an intensity score from 0(none) to 5(worst). Therefore, the suicidal ideation intensity total score range from 0 to 25, with a score of 0 given for no suicidal ideation.
Time Frame: Da y 1, Da y 6, Day 30, Day 60, Day 90 and Day 180
Population: Safety Population. Number of participants with at least one on-treatment C-SSRS assessment were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo - Safety | GSK249320 15 mg/kg - Safety
Number analyzed (Participants) | 63 | 63
Participants | 10 | 3

22. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for GSK249320
Description: Cmax is the maximum observed concentration of GSK249320 obtained at the end of infusion post dose on Day 6. Due to early termination of the study, this data was not collected.
Time Frame: Pre-dose and post-dose up to Day 180
Population: The Pharmacokinetics (PK) population consisted of all participants in the Safety population who have at least one PK sample with a concentration above the non-quantifiable limit. Data not collected due to early termination of study.
Groups:
- GSK249320 15 mg/kg - PK: Participants received GSK249320 15 mg/kg administered as two IV infusions, the first on Study Day 1 which is 24-72 post-stroke onset, and the second on Study Day 6 (+/- 2 days). Each 100 mL IV infusion was delivered over a period of 75 minutes (a 60 minute infusion followed by a 10 to 15 minute flush). PK population consisted of all participants in the Safety population who have at least one PK sample with a concentration above the non-quantifiable limit.
Arm/Group | GSK249320 15 mg/kg - PK
Number analyzed (Participants) | 0

23. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) GSK249320
Description: Tmax is the time of the occurrence of Cmax. The Cmax is defined as the maximum observed concentration of GSK249320 obtained at the end of infusion post dose on day 6. Due to early termination of the study data for Tmax was not collected.
Time Frame: Pre-dose and post-dose up to Day 180
Population: PK population. Due to early termination of the study, data for Tmax was not collected
Arm/Group | GSK249320 15 mg/kg - PK
Number analyzed (Participants) | 0

24. Secondary Outcome: PK as Measured by Plasma Decay Half-life (t1/2) GSK249320
Description: Blood samples were collected for determination of plasma concentrations of GSK249320. Terminal phase half-life was derived from the plasma concentration-time data. Only participants in the GSK249320 15 mg/kg group were analyzed.
Time Frame: Up to Day 180
Population: PK Population.
Measure: Median (Full Range); unit: Days
Groups:
- GSK249320 15 mg/kg - PK: Participants received GSK249320 15 mg/kg administered as two IV infusions, the first on Study Day 1 which is 24-72 post-stroke onset, and the second on Study Day 6 (+/- 2 days). Each 100 mL IV infusion was delivered over a period of 75 minutes (a 60 minute infusion followed by a 10 to 15 minute flush).
Arm/Group | GSK249320 15 mg/kg - PK
Number analyzed (Participants) | 62
Days | 23.09 [13.5 to 42.9]

25. Secondary Outcome: Area Under the Concentration-time Curve From 0 to 5 Days [AUC(0-5d)] and Area Under the Concentration-time Curve From Time Zero (Pre-dose) Extrapolated to Infinite Time [AUC(0-inf)] for GSK249320
Description: Blood samples were collected for determination of plasma concentrations of GSK249320. AUC (0-5d) and AUC (0-inf) were derived from the plasma concentration-time data. AUC(0-5d) is the model predicted AUC over the planned TAU of 5 days. Only participants in the GSK249320 15 mg/kg group were analyzed.
Time Frame: Pre-dose and post-dose up to Day 180
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligrams/milliliter*hour
Arm/Group | GSK249320 15 mg/kg - PK
Number analyzed (Participants) | 62
Milligrams/milliliter*hour
  AUC(0-5 d) | 28.2273 (10.9)
  AUC(0-inf) | 120.6895 (20.4)

26. Secondary Outcome: Clearance (CL) for GSK249320
Description: Blood samples were collected for determination of plasma concentrations of GSK249320. CL was derived from the plasma concentration-time data. Analysis was performed for PK Population that comprised of all participants in the Safety Population who had at least one PK sample with a concentration above the non-quantifiable limit. Only participants in the GSK249320 15 mg/kg group were analyzed.
Time Frame: Up to Day 180
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligrams/kilograms/hour
Arm/Group | GSK249320 15 mg/kg - PK
Number analyzed (Participants) | 62
Milligrams/kilograms/hour | 0.1243 (20.4)

27. Secondary Outcome: Volume of Distribution (V1 and V2) and Volume at Steady State (Vss) for GSK249320
Description: Blood samples were collected for determination of plasma concentrations of GSK249320. V1, V2 and Vss were derived from the plasma concentration-time data. Analysis was performed for PK Population that comprised of all participants in the Safety Population who had at least one PK sample with a concentration above the non-quantifiable limit. Only participants in the GSK249320 15 mg/kg group were analyzed.
Time Frame: Up to Day 180
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliters/kilogram
Groups:
- GSK249320 15 mg/kg - PK: Participants received GSK249320 15 mg/kg, administered as two IV infusions, the first on Study Day 1 which is 24-72 post-stroke onset, and the second on Study Day 6 (+/- 2 days). Each 100 mL IV infusion was delivered over a period of 75 minutes (a 60 minute infusion followed by a 10 to 15 minute flush). PK population consisted of all participants in the Safety population who have at least one PK sample with a concentration above the non-quantifiable limit.
Arm/Group | GSK249320 15 mg/kg - PK
Number analyzed (Participants) | 62
milliliters/kilogram
  V1 | 43.6992 (6.7)
  V2 | 41.4193 (17.8)
  Vss | 85.2892 (11.5)

28. Secondary Outcome: Antibodies Against GSK249320, Assessed Using Electrochemi-luminescent Assay (ECL) Assay
Description: Blood samples were collected and the presence of antibodies against GSK249320 was assessed using ECL assays. Positive result indicated presence of antibodies and negative result indicated absence of antibodies. Confirmed samples with presence of antibodies were further characterized for neutralizing activity as binding antibody (BAb) and neutralising antibody (NAb) by a neutralization assay.By-visit sample sizes vary due to missing data or early termination of the study.
Time Frame: Day 1, Day 30, Day 180, EW visit and Follow-up visit
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo - Safety | GSK249320 15 mg/kg - Safety
Number analyzed (Participants) | 68 | 65
Participants
  Day 1, BAb Positive | 7 | 5
  Day 1, BAb Negative | 60 | 59
  Day 1, NAb Negative: number analyzed (Participants) | 7 | 5
  Day 1, NAb Negative | 0 | 2
  Day 30, BAb Positive: number analyzed (Participants) | 59 | 60
  Day 30, BAb Positive | 4 | 4
  Day 30, BAb Negative: number analyzed (Participants) | 59 | 60
  Day 30, BAb Negative | 44 | 46
  Day 30, NAb Negative: number analyzed (Participants) | 4 | 4
  Day 30, NAb Negative | 1 | 1
  Day 180, BAb Positive: number analyzed (Participants) | 42 | 41
  Day 180, BAb Positive | 0 | 5
  Day 180, BAb Negative: number analyzed (Participants) | 42 | 41
  Day 180, BAb Negative | 24 | 19
  EW visit, BAb Positive: number analyzed (Participants) | 23 | 23
  EW visit, BAb Positive | 1 | 4
  EW visit, BAb Negative: number analyzed (Participants) | 23 | 23
  EW visit, BAb Negative | 22 | 18
  EW visit, NAb Negative: number analyzed (Participants) | 1 | 4
  EW visit, NAb Negative | 1 | 4
  FU visit, BAb Positive: number analyzed (Participants) | 0 | 1
  FU visit, BAb Positive | 0 | 1
  FU visit, NAb Negative: number analyzed (Participants) | 0 | 1
  FU visit, NAb Negative | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 14 months
Description: SAEs and non-serious AEs were reported for members of the Safety Population, comprised of all participants who were randomized and took at least one dose of study medication.
Groups:
- Placebo: Participants received placebo administered as two IV infusions, the first on Study Day 1 which is 24-72 hours post-stroke onset, and the second on Study Day 6 (+/- 2 days). Each 100 mL, IV infusion was delivered over a period of 75 minutes (a 60 minute infusion followed by a 10 to 15 minute flush).
Arm/Group | Placebo | GSK249320 15 mg/kg
All-Cause Mortality (participants affected / at risk) | 5/68 | 2/65
Serious Adverse Events (participants affected / at risk) | 16/68 | 9/65
Other Adverse Events (participants affected / at risk) | 25/68 | 32/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=68) | GSK249320 15 mg/kg (N=65)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 0 | 1
Anal ulcer (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Brain edema (Nervous system disorders) | 1 | 0
Cerebral hemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Haemorrhagic transformation stroke (Nervous system disorders) | 0 | 1
Ischemic cerebral infarction (Nervous system disorders) | 0 | 1
Stroke in evolution (Nervous system disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Neck injury (Injury, poisoning and procedural complications) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1
Hypertensive emergency (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=68) | GSK249320 15 mg/kg (N=65)
Hypertension (Vascular disorders) | 4 | 3
Hypotension (Vascular disorders) | 4 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 4
Headache (Nervous system disorders) | 7 | 12
Insomnia (Psychiatric disorders) | 4 | 5
Constipation (Gastrointestinal disorders) | 6 | 13
Nausea (Gastrointestinal disorders) | 3 | 5
Rash (Skin and subcutaneous tissue disorders) | 3 | 4
Urinary tract infection (Gastrointestinal disorders) | 4 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early, on 27 May 2014, at the planned interim analysis for futility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.